CLINICAL TRIAL: NCT01526629
Title: Identification of Implantable Cardioverter Defibrillator Patients With Remote Follow up That Requires an Onsite Visit
Brief Title: Full Automaticity and Remote Follow-up
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 1047
Record Dates: First submitted 2011-11-14; First posted 2012-02-06 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2017-02

CONDITIONS: Tachyarrhythmia
Keywords: ICD; Remote follow-up
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD patients with remote follow-up: Patients implanted with a fully automatic ICD and remotely followed-up.

SUMMARY:
With the expansion of Sudden Cardiac Death (SCD) primary prevention indications, the number of Implantable Cardioverter Defibrillators (ICD) implants has increased significantly in the recent years. This has resulted in an increase of the number of follow-up (FU) to be performed and a growing workload for centers. Remote FU system such as the Medtronic Carelink system allows to check remotely the proper functioning of self evaluating devices and give informations of some clinical events.

The objective of this study is to define which patients with a remote follow-up need additional onsite visit and to assess to which extent remote FU can be an alternative to onsite visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18,
* Patient implanted with a fully automatic ICD and remotely followed-up,
* Patient geographically stable and able to attend FU at investigative site
* Patient who signed a data release authorization form,

Exclusion Criteria:

* Patient whose mental or physical capacity impedes to give an informed data release authorization,
* Patient already enrolled in a clinical study whose procedures may interfere with the results of the present study,
* Patients in New York Heart Association (NYHA) class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient implanted with a sigle- or dual-chamber ICD or a Cardiac Resynchronization-Defibrillator system (CRT-D) and remotely followed-up
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walid Amara, MD, Principal Investigator — Centre Hospitalier de Montfermeil
Locations (1):
- CH Montfermeil, Montfermeil, France

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICD Patients With Remote Follow-up
Started | 354
Completed | 308
Not Completed | 46

BASELINE CHARACTERISTICS:
Arm/Group | ICD Patients With Remote Follow-up
Number analyzed (Participants) | 354
Age, Customized [Mean (Full Range); unit: years]
  Men | 65 [55 to 75]
  Women | 56 [42 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 288
Region of Enrollment [Number; unit: participants]
  France | 354

OUTCOME MEASURES:

1. Primary Outcome: Remote Follow-up as an Alternative to Onsite Visit
Description: Evaluate the percentage of patients who had a successful remote follow up, as an alternative to onsite visit for patients implanted with a fully automatic ICD
Time Frame: 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | ICD Patients With Remote Follow-up
Number analyzed (Participants) | 308
Participants | 203

ADVERSE EVENTS:
Arm/Group | ICD Patients With Remote Follow-up
Serious Adverse Events (participants affected / at risk) | 75/354
Other Adverse Events (participants affected / at risk) | 0/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ICD Patients With Remote Follow-up (N=354)
Death (General disorders) | 10
Ventricular arrhytmias (Cardiac disorders) | 9
Cardiac decompensation (Cardiac disorders) | 14
Atrial arrhytmias (Cardiac disorders) | 6
Infection or pocket hematoma (Skin and subcutaneous tissue disorders) | 5
Event of aggravation (Cardiac disorders) | 6 — dyspnea, heart failure, stroke...
cardiovascular procedures (Cardiac disorders) | 4 — stent, ablation, transplantation..;
cardiovascular complication (Cardiac disorders) | 5 — aneurysm, pericarditis, stenosis...
Non cardiovascular causes (General disorders) | 12
Integrity default of material components (Injury, poisoning and procedural complications) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No